CLINICAL TRIAL: NCT00661973
Title: The Effect of Inhaled Corticosteroids (ICS) on Airway Smooth Muscle in Asthma
Brief Title: Inhaled Corticosteroids on Airway Smooth Muscle in Asthma
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn for administrative reasons
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2007-006664-29; 07/H0803/239
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Asthma
Keywords: asthma; airway smooth muscle; inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- overall (Experimental)
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — inhaled budesonide (turbohaler) 400 micrograms twice a day for 4 weeks
  Other Names: pulmicort

SUMMARY:
The main objective is to evaluate how treatment with inhaled corticosteroids (ICS) affects the characteristics of airway smooth muscle (ASM) cells from asthmatic subjects. Our hypothesis is that airway smooth muscle cell dysfunction plays an important role in the pathogenesis of asthma, and that treatment with inhaled corticosteroids reverses the abnormalities in airway smooth muscle cell function.

DETAILED DESCRIPTION:
Aims and Objectives

Most of the work published to date on the effect of steroids on ASM has been carried out in animal models or in in vitro experiments. We would like to evaluate in vivo whether abnormalities in ASM function respond to ICS. Because ASM cells can be obtained from bronchial biopsies obtained via bronchoscopy, we will examine endobronchial biopsies from corticosteroid-naïve, mild asthmatic subjects. In particular, we will examine whether ICS have any effect ASM mass, proliferation and expression of different contractile proteins (α-actin and myosin) and chemokines, and will assess in vitro the response of ASM cells to stimulation by TGF-β and IL-1β. We will also examine the effect of dexamethasone on chemokine release and induced proliferation in vitro before and after treatment with ICS.

We will examine the effect of inhaled corticosteroids in 12 subjects with mild asthma. The subjects will be studied during a baseline period and again after receiving treatment with inhaled corticosteroid therapy with Budesonide Turbohaler (400 ug bd) for 4 weeks. The results of these two periods will be compared.

There will be 5 study visits. In the first two visits, the subjects will undergo spirometry with reversibility testing, a methacholine challenge test, skin prick tests and IgE levels, measurement of exhaled nitric oxide, and subjects will complete an Asthma Control Questionnaire and an Asthma Quality of Life Questionnaire. The third visit will be the day admission for the bronchoscopy. They will be given asthma control diary cards to complete during the 4-week treatment with ICS and receive their ICS turbohaler. At visit 4, they will have repeat spirometry and methacholine challenge to assess if there has been a change secondary to treatment with ICS. The final visit will be for the second bronchoscopy, when the dairy card and ICS inhaler will be collected, and the subjects will complete the Asthma Control and Quality of Life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of asthma
* Age 18-60
* Intermittent asthma symptoms < once/week
* FEV1>80% of predicted
* Not on inhaled corticosteroid therapy

Exclusion Criteria:

* Previous long-term use of inhaled corticosteroids (within 1 year of entry into study)
* Past history of hypersensitivity to budesonide
* Current smokers, or less than 3 years since quitting smoking
* Less than 4 weeks from an exacerbation
* On steroid-sparing agent or immunosuppressant such as azathioprine, methotrexate and ciclosporin
* Concomitant anti-IgE therapy
* Pregnancy
* Previous bronchoscopy within three months of this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Changes in ASM mass, proliferation and migration after ICS therapy; changes in chemokine release after ICS therapy | 4 weeks

SECONDARY OUTCOMES:
Changes in sub-basement membrane thickness and inflammatory cell count after ICS therapy | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kian F Chung, MBBS FRCP MD DSc, Principal Investigator — Imperial College London
Locations (1):
- Asthma lab, Royal Brompton Hospital, Sydney Street, London, United Kingdom